CLINICAL TRIAL: NCT02174081
Title: ARDS Prediction Score in Critically Ill Patients in China
Status: Completed | Type: Observational
Sponsor: Jianfeng Xie (Other)
Responsible Party: Sponsor-Investigator, Jianfeng Xie, Zhongda Hospital, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: ARDS Prediction system
Record Dates: First submitted 2014-06-11; First posted 2014-06-25 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: ARDS; Septic Shock
Keywords: mechanical ventilation, ARDS, Ventilator strategy, outcome
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
ARDS is a severe disease, it's important to predict the incidence of ARDS.

DETAILED DESCRIPTION:
From January 1 to January 31, 2012 and from January 1 to January 10, 2013 , all patients admit to the ICUs will be enrolled. The demographic characteristics, diagnosis, formerly medical history, Ventilator indications, Ventilator data, other respiratory treatments, weaning outcome and 28 day mortality will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Critically ill patients who admitted into participating ICU

Exclusion Criteria:

Patients with chronic pulmonary disease such as chronic obstructive pulmonary disease (COPD), asthma, lung cancer, pulmonary fibrosis and tuberculosis Age less than 18 years old Pregnancy Died within 24 hours from ICU admission ARDS patients who diagnosed 24hours before ICU admission Referral from other hospital to participating ICU Lack of data of ARDS risk factors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients have the risk of ARDS
Sampling Method: Probability Sample
Enrollment: 698 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
incidence of ARDS | up to 24 months
  evaluate the incidence of risk factors of ARDS

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Xie, Dr, Principal Investigator — Southeast University
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China